CLINICAL TRIAL: NCT06357286
Title: Unstable Income, Rising Stress? The Effect of Income Instability on Psychological and Physiological Health, Pilot Study
Brief Title: Income Volatility and Mental Health, Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB0148156
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): The Control arm will not be hired by the cash-for-work program but will be surveyed.
- Stable income arm (Experimental): The Stable Income arm will work the same number of hours (36) and earn the same amount (108 cedis) every period.
  Interventions: Behavioral: Work opportunities
- Predictable Instability Arm (Experimental): The hours and earnings of the Predictable Instability arm will vary over time. In three periods, the participant will work longer hours (60) and will earn more (180 cedis). In the remaining three periods, she will work fewer hours (12) and will earn less (36 cedis). Crucially, she will be able to predict all swings in her study earnings in the future-i.e., she will know her hours and earnings in each future period.
  Interventions: Behavioral: Work opportunities
- Unpredictable Instability Arm (Experimental): The hours and earnings of the Unpredictable Instability arm will vary unpredictably over time. In any given period, there will be a 50% chance that she works longer hours (60) and earns more (180 cedis) and a 50% chance that she works fewer hours (12) and earns less (36 cedis).
  Interventions: Behavioral: Work opportunities

INTERVENTIONS:
Behavioral: Work opportunities — Individuals in the treated arms of the study will be offered work opportunities (sewing bags) to earn cash. The timing of these opportunities and knowledge of the amount and timing varies by experimental arm.
  Arms: Predictable Instability Arm; Stable income arm; Unpredictable Instability Arm

SUMMARY:
Income instability is a defining aspect of the lives of the poor, who also disproportionately suffer from poor mental and physical health. Our research is the first to assess the causal effects of predictable and unpredictable income instability on the psychological and physical health of the poor. It will advance the scientific knowledge on the effects of economic instability as well as our understanding of health disparities.

DETAILED DESCRIPTION:
The poor suffer disproportionally from poor mental and physical health. Many causes for these disparities have been considered, including low income. But, poor families' incomes are not only low, but also often unstable and unpredictable. This instability creates uncertainty about whether they will be able to safeguard their future wellbeing. According to the allostatic load framework, prolonged activation of physiological stress responses will cause "wear and tear" on the body, heightening risks of cardiovascular disease and of age-related metabolic diseases, promoting cognitive decline and dementia, and accelerating cellular aging.

This research will study the causal effects of income instability on the psychological and physical health of the poor. Our specific aims are to: 1) Identify the causal effect of income instability on psychological health (e.g. depression, anxiety), biomarkers of stress (e.g. cortisol), and physical health (e.g. blood pressure), 2) Decompose the effects identified in aim 1 into the effects of predictable and unpredictable instability and compare to the impact of increasing the average level of income, and 3) Investigate the channels through which effects on health occur, including both economic and behavioral channels and estimate the impact of key moderating factors (e.g. age, gender, baseline mental health).

The trial will be conducted in northern Ghana. We will manipulate income instability by varying the number of work hours (and hence earnings) of participants in a cash-for-work program. Participants in the first treatment arm will have a fixed work schedule, with the same hours and earning each period. The hours and earnings of a second treatment arm will vary over time, but the fluctuations will be known in advance. Finally, the number of work hours and earnings of a third treatment arm will fluctuate unpredictably. Each of these arms will be compared to a control group that is surveyed, but not offered additional work. Importantly, we will vary income instability while holding the average level of income constant in order to disentangle the impact of instability from the level-effect.

The full study will create 1,867 new jobs that would not otherwise be available during the lean season when jobs are scarce. The intervention has been designed so that the job opportunity cannot make them worse off than they would otherwise have been in the absence of research.

Please note this registration is for a pilot study (n= approximately 400) prior to the main experiment. As such, we anticipate the pilot will be underpowered and do not expect to find significant effects.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 65
* female
* lives in a household with fewer than 5 adults

Exclusion Criteria:

* Pregnancy at enrollment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2024-05-25 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Innovations for Poverty Action, Tamale, Ghana

IPD SHARING:
Plan to Share IPD: Undecided
De-identified survey data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Stable Income Arm | Predictable Instability Arm | Unpredictable Instability Arm
Started | 70 | 80 | 83 | 157
Completed | 67 | 80 | 82 | 155
Not Completed | 3 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Stable Income Arm | Predictable Instability Arm | Unpredictable Instability Arm | Total
Number analyzed (Participants) | 70 | 80 | 83 | 157 | 390
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 70 | 80 | 83 | 157 | 390
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (10.9) | 36.5 (10.4) | 37.2 (11.4) | 37.7 (11.8) | 37.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 80 | 83 | 157 | 390
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 70 | 80 | 83 | 157 | 390
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Ghana | 70 | 80 | 83 | 157 | 390

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: Patient Health Questionnaire (PHQ)-8, each item is scored 0-3. Multiplying the range per item (0-3) by the number of items (8) gives the total corresponding range of the scale: 0 to 24. Higher scores indicate worse mental health.
Time Frame: The measurement was taken at endline (after 8 weeks of intervention). Respondents were asked to evaluate each item over the last two weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Stable Income Arm | Predictable Instability Arm | Unpredictable Instability Arm
Number analyzed (Participants) | 67 | 80 | 82 | 155
units on a scale | 7.4 (4.4) | 5.7 (4.1) | 6.3 (4.0) | 7.4 (4.8)

ADVERSE EVENTS:
Time Frame: 4 months
Description: Follow standard definitions
Arm/Group | Control | Stable Income Arm | Predictable Instability Arm | Unpredictable Instability Arm
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/80 | 0/83 | 0/157
Serious Adverse Events (participants affected / at risk) | 3/70 | 0/80 | 0/83 | 2/157
Other Adverse Events (participants affected / at risk) | 13/70 | 21/80 | 29/83 | 52/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=70) | Stable Income Arm (N=80) | Predictable Instability Arm (N=83) | Unpredictable Instability Arm (N=157)
hospitalized for fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Participant was hospitalized for fever (e.g. malaria, other infectious disease)
pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — participant fell while carrying water and sustained an injury
pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant experienced severe stomach pains
pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — participant experienced severe leg pain
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=70) | Stable Income Arm (N=80) | Predictable Instability Arm (N=83) | Unpredictable Instability Arm (N=157)
accidents and injuries (General disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4) — accidents (i.e. road traffic) and injuries (i.e. cutting oneself with a knife)
pain (General disorders) | 6 (7) | 1 (1) | 4 (4) | 13 (13) — pain of any body part other than the head
fatigue and/or dizziness (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) — fatigue and/or dizziness
gastrointestinal distress (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3) | 5 (5) — gastrointestinal distress (i.e. stomachache, vomiting, diarrhea)
headache (General disorders) | 2 (2) | 5 (5) | 5 (6) | 8 (8) — headache
infectious diseases (Infections and infestations) | 3 (3) | 7 (7) | 13 (14) | 20 (23) — malaria, fever, etc
rash or swelling (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — rash or swelling
spiritual illness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — possession, feelings of malaise

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT06357286/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT06357286/ICF_001.pdf